CLINICAL TRIAL: NCT03011138
Title: The Relationship Between Gait Velocity and Gait Parameters
Status: Completed | Type: Observational
Sponsor: Guangzhou General Hospital of Guangzhou Military Command (Other)
Collaborators: Medical Center of Assessment, Prevention and Treatment of Bone & Joint Diseases, Guangdong, China (Other); The First Affiliated Hospital of Guangzhou Medical University (Other)
Responsible Party: Principal Investigator, Yu Zhang, chief surgeon, associate professor, Guangzhou General Hospital of Guangzhou Military Command
Other Study IDs: GuangzhouGH004
Record Dates: First submitted 2017-01-03; First posted 2017-01-05 (Estimated); Last update posted 2017-02-13 (Actual); Status verified 2017-02

CONDITIONS: Gait Velocity
Keywords: knee; gait velocity; kinematic parameters

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (7):
- V 1: Gait velocity will be set at 1.0km/h.
  Interventions: Procedure: Gait velocity
- V 2: Gait velocity will be set at 1.5km/h.
  Interventions: Procedure: Gait velocity
- V 3: Gait velocity will be set at 2.0km/h.
  Interventions: Procedure: Gait velocity
- V 4: Gait velocity will be set at 2.5km/h.
  Interventions: Procedure: Gait velocity
- V 5: Gait velocity will be set at 3.0km/h.
  Interventions: Procedure: Gait velocity
- V 6: Gait velocity will be set at 3.5km/h.
  Interventions: Procedure: Gait velocity
- V 7: Gait velocity will be set at 4.0km/h.
  Interventions: Procedure: Gait velocity

INTERVENTIONS:
Procedure: Gait velocity — Once participants are eligible, they will undergo the experimental procedure. Before data collection, they will walk on a treadmill in barefoot for ten minutes to adapt the condition. The a gait analysis system will collect the data while they walk on the treadmill in barefoot at selected gait speed.

SUMMARY:
Previous reports have the evidence implicating gait velocity may affect kinematic parameters. However, how the gait velocity will influence kinematic parameters remain unclear. The purpose of this research is to find out kinematic characteristics among different gait velocity. To do this, it will provide a reference for future prospective studies or investigations and make us fully understand the impact of gait velocity.

ELIGIBILITY:
Inclusion Criteria:

1. 20< age < 30.
2. Body mass index < 30.
3. No history of major injury or surgery in lower limbs.
4. No symptoms of lower limbs.
5. Physical examination to test the lower limbs to be normal.
6. The habit of moderate exercise (e.g. Jogging) at least once a week for at least 30 minutes.

Exclusion Criteria:

1. Body mass index >30.
2. Injury or surgery in hip/knee/ankle.
3. History trauma in the lower limbs (e.g. fracture).
4. Neuropathic disease.
5. Muscular disease.
6. Lack ability to finish the procedure physically or mentally.
7. Easy to fall.
8. Any other conditions that can influence gait parameters of the lower limbs.

Ages: 20 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: All the participants will be recruited via university advertisement.
Sampling Method: Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2017-01-01 (Actual); Primary Completion 2017-02-01 (Actual); Study Completion 2017-02-06 (Actual)

PRIMARY OUTCOMES:
Knee flexion/extension angle at initial contact during gait. | 1 Day
  The gait cycle include seven key events (e.g. initial contact), and each gait has six degrees of freedom, including knee flexion/extension, internal/external rotation, adduction/abduction, anterior/posterior translation, distal/proximal translation, medial/lateral translation. The unit of angle is degree and that of translation is millimetre.
Knee internal/external rotation angle at initial contact during gait. | 1 Day
  The gait cycle include seven key events (e.g. initial contact), and each gait has six degrees of freedom, including knee flexion/extension, internal/external rotation, adduction/abduction, anterior/posterior translation, distal/proximal translation, medial/lateral translation. The unit of angle is degree and that of translation is millimetre.
Knee adduction/abduction angle at initial contact during gait. | 1 Day
  The gait cycle include seven key events (e.g. initial contact), and each gait has six degrees of freedom, including knee flexion/extension, internal/external rotation, adduction/abduction, anterior/posterior translation, distal/proximal translation, medial/lateral translation. The unit of angle is degree and that of translation is millimetre.
Knee anterior/posterior translation at initial contact during gait. | 1 Day
  The gait cycle include seven key events (e.g. initial contact), and each gait has six degrees of freedom, including knee flexion/extension, internal/external rotation, adduction/abduction, anterior/posterior translation, distal/proximal translation, medial/lateral translation. The unit of angle is degree and that of translation is millimetre.
Knee medial/lateral translation at initial contact during gait. | 1 Day
  The gait cycle include seven key events (e.g. initial contact), and each gait has six degrees of freedom, including knee flexion/extension, internal/external rotation, adduction/abduction, anterior/posterior translation, distal/proximal translation, medial/lateral translation. The unit of angle is degree and that of translation is millimetre.
Knee proximal/distal translation at initial contact during gait. | 1 Day
  The gait cycle include seven key events (e.g. initial contact), and each gait has six degrees of freedom, including knee flexion/extension, internal/external rotation, adduction/abduction, anterior/posterior translation, distal/proximal translation, medial/lateral translation. The unit of angle is degree and that of translation is millimetre.
Knee flexion/extension angle at opposite toe off during gait. | 1 Day
  The gait cycle include seven key events (e.g. initial contact), and each gait has six degrees of freedom, including knee flexion/extension, internal/external rotation, adduction/abduction, anterior/posterior translation, distal/proximal translation, medial/lateral translation. The unit of angle is degree and that of translation is millimetre.
Knee adduction/abduction angle at opposite toe off during gait. | 1 Day
  The gait cycle include seven key events (e.g. initial contact), and each gait has six degrees of freedom, including knee flexion/extension, internal/external rotation, adduction/abduction, anterior/posterior translation, distal/proximal translation, medial/lateral translation. The unit of angle is degree and that of translation is millimetre.
Knee internal/external rotation angle at opposite toe off during gait. | 1 Day
  The gait cycle include seven key events (e.g. initial contact), and each gait has six degrees of freedom, including knee flexion/extension, internal/external rotation, adduction/abduction, anterior/posterior translation, distal/proximal translation, medial/lateral translation. The unit of angle is degree and that of translation is millimetre.
Knee anterior/posterior translation at opposite toe off during gait. | 1 Day
  The gait cycle include seven key events (e.g. initial contact), and each gait has six degrees of freedom, including knee flexion/extension, internal/external rotation, adduction/abduction, anterior/posterior translation, distal/proximal translation, medial/lateral translation. The unit of angle is degree and that of translation is millimetre.
Knee distal/proximal translation at opposite toe off during gait. | 1 Day
  The gait cycle include seven key events (e.g. initial contact), and each gait has six degrees of freedom, including knee flexion/extension, internal/external rotation, adduction/abduction, anterior/posterior translation, distal/proximal translation, medial/lateral translation. The unit of angle is degree and that of translation is millimetre.
Knee medial/lateral translation at opposite toe off during gait. | 1 Day
  The gait cycle include seven key events (e.g. initial contact), and each gait has six degrees of freedom, including knee flexion/extension, internal/external rotation, adduction/abduction, anterior/posterior translation, distal/proximal translation, medial/lateral translation. The unit of angle is degree and that of translation is millimetre.
Knee flexion/extension angle at heel rise during gait. | 1 Day
  The gait cycle include seven key events (e.g. initial contact), and each gait has six degrees of freedom, including knee flexion/extension, internal/external rotation, adduction/abduction, anterior/posterior translation, distal/proximal translation, medial/lateral translation. The unit of angle is degree and that of translation is millimetre.
Knee internal/external rotation angle at heel rise during gait. | 1 Day
  The gait cycle include seven key events (e.g. initial contact), and each gait has six degrees of freedom, including knee flexion/extension, internal/external rotation, adduction/abduction, anterior/posterior translation, distal/proximal translation, medial/lateral translation. The unit of angle is degree and that of translation is millimetre.
Knee adduction/abduction angle at heel rise during gait. | 1 Day
  The gait cycle include seven key events (e.g. initial contact), and each gait has six degrees of freedom, including knee flexion/extension, internal/external rotation, adduction/abduction, anterior/posterior translation, distal/proximal translation, medial/lateral translation. The unit of angle is degree and that of translation is millimetre.
Knee anterior/posterior translation at heel rise during gait. | 1 Day
  The gait cycle include seven key events (e.g. initial contact), and each gait has six degrees of freedom, including knee flexion/extension, internal/external rotation, adduction/abduction, anterior/posterior translation, distal/proximal translation, medial/lateral translation. The unit of angle is degree and that of translation is millimetre.
Knee distal/proximal translation at heel rise during gait. | 1 Day
  The gait cycle include seven key events (e.g. initial contact), and each gait has six degrees of freedom, including knee flexion/extension, internal/external rotation, adduction/abduction, anterior/posterior translation, distal/proximal translation, medial/lateral translation. The unit of angle is degree and that of translation is millimetre.
Knee medial/lateral translation at heel rise during gait. | 1 Day
  The gait cycle include seven key events (e.g. initial contact), and each gait has six degrees of freedom, including knee flexion/extension, internal/external rotation, adduction/abduction, anterior/posterior translation, distal/proximal translation, medial/lateral translation. The unit of angle is degree and that of translation is millimetre.
Knee flexion/extension angle at opposite initial contact during gait. | 1 Day
  The gait cycle include seven key events (e.g. initial contact), and each gait has six degrees of freedom, including knee flexion/extension, internal/external rotation, adduction/abduction, anterior/posterior translation, distal/proximal translation, medial/lateral translation. The unit of angle is degree and that of translation is millimetre.
Knee adduction/abduction angle at opposite initial contact during gait. | 1 Day
  The gait cycle include seven key events (e.g. initial contact), and each gait has six degrees of freedom, including knee flexion/extension, internal/external rotation, adduction/abduction, anterior/posterior translation, distal/proximal translation, medial/lateral translation. The unit of angle is degree and that of translation is millimetre.
Knee internal/external rotation angle at opposite initial contact during gait. | 1 Day
  The gait cycle include seven key events (e.g. initial contact), and each gait has six degrees of freedom, including knee flexion/extension, internal/external rotation, adduction/abduction, anterior/posterior translation, distal/proximal translation, medial/lateral translation. The unit of angle is degree and that of translation is millimetre.
Knee anterior/posterior translation at opposite initial contact during gait. | 1 Day
  The gait cycle include seven key events (e.g. initial contact), and each gait has six degrees of freedom, including knee flexion/extension, internal/external rotation, adduction/abduction, anterior/posterior translation, distal/proximal translation, medial/lateral translation. The unit of angle is degree and that of translation is millimetre.
Knee distal/proximal translation at opposite initial contact during gait. | 1 Day
  The gait cycle include seven key events (e.g. initial contact), and each gait has six degrees of freedom, including knee flexion/extension, internal/external rotation, adduction/abduction, anterior/posterior translation, distal/proximal translation, medial/lateral translation. The unit of angle is degree and that of translation is millimetre.
Knee medial/lateral translation at opposite initial contact during gait. | 1 Day
  The gait cycle include seven key events (e.g. initial contact), and each gait has six degrees of freedom, including knee flexion/extension, internal/external rotation, adduction/abduction, anterior/posterior translation, distal/proximal translation, medial/lateral translation. The unit of angle is degree and that of translation is millimetre.
Knee flexion/extension angle at toe off during gait. | 1 Day
  The gait cycle include seven key events (e.g. initial contact), and each gait has six degrees of freedom, including knee flexion/extension, internal/external rotation, adduction/abduction, anterior/posterior translation, distal/proximal translation, medial/lateral translation. The unit of angle is degree and that of translation is millimetre.
Knee adduction/abduction angle at toe off during gait. | 1 Day
  The gait cycle include seven key events (e.g. initial contact), and each gait has six degrees of freedom, including knee flexion/extension, internal/external rotation, adduction/abduction, anterior/posterior translation, distal/proximal translation, medial/lateral translation. The unit of angle is degree and that of translation is millimetre.
Knee internal/external rotation angle at toe off during gait. | 1 Day
  The gait cycle include seven key events (e.g. initial contact), and each gait has six degrees of freedom, including knee flexion/extension, internal/external rotation, adduction/abduction, anterior/posterior translation, distal/proximal translation, medial/lateral translation. The unit of angle is degree and that of translation is millimetre.
Knee anterior/posterior translation at toe off during gait. | 1 Day
  The gait cycle include seven key events (e.g. initial contact), and each gait has six degrees of freedom, including knee flexion/extension, internal/external rotation, adduction/abduction, anterior/posterior translation, distal/proximal translation, medial/lateral translation. The unit of angle is degree and that of translation is millimetre.
Knee distal/proximal translation at toe off during gait. | 1 Day
  The gait cycle include seven key events (e.g. initial contact), and each gait has six degrees of freedom, including knee flexion/extension, internal/external rotation, adduction/abduction, anterior/posterior translation, distal/proximal translation, medial/lateral translation. The unit of angle is degree and that of translation is millimetre.
Knee medial/lateral translation at toe off during gait. | 1 Day
  The gait cycle include seven key events (e.g. initial contact), and each gait has six degrees of freedom, including knee flexion/extension, internal/external rotation, adduction/abduction, anterior/posterior translation, distal/proximal translation, medial/lateral translation. The unit of angle is degree and that of translation is millimetre.
Knee flexion/extension angle at feet adjacent during gait. | 1 Day
  The gait cycle include seven key events (e.g. initial contact), and each gait has six degrees of freedom, including knee flexion/extension, internal/external rotation, adduction/abduction, anterior/posterior translation, distal/proximal translation, medial/lateral translation. The unit of angle is degree and that of translation is millimetre.
Knee internal/external rotation angle at feet adjacent during gait. | 1 Day
  The gait cycle include seven key events (e.g. initial contact), and each gait has six degrees of freedom, including knee flexion/extension, internal/external rotation, adduction/abduction, anterior/posterior translation, distal/proximal translation, medial/lateral translation. The unit of angle is degree and that of translation is millimetre.
Knee adduction/abduction angle at feet adjacent during gait. | 1 Day
  The gait cycle include seven key events (e.g. initial contact), and each gait has six degrees of freedom, including knee flexion/extension, internal/external rotation, adduction/abduction, anterior/posterior translation, distal/proximal translation, medial/lateral translation. The unit of angle is degree and that of translation is millimetre.
Knee anterior/posterior translation at feet adjacent during gait. | 1 Day
  The gait cycle include seven key events (e.g. initial contact), and each gait has six degrees of freedom, including knee flexion/extension, internal/external rotation, adduction/abduction, anterior/posterior translation, distal/proximal translation, medial/lateral translation. The unit of angle is degree and that of translation is millimetre.
Knee distal/proximal translation at feet adjacent during gait. | 1 Day
  The gait cycle include seven key events (e.g. initial contact), and each gait has six degrees of freedom, including knee flexion/extension, internal/external rotation, adduction/abduction, anterior/posterior translation, distal/proximal translation, medial/lateral translation. The unit of angle is degree and that of translation is millimetre.
Knee medial/lateral translation at feet adjacent during gait. | 1 Day
  The gait cycle include seven key events (e.g. initial contact), and each gait has six degrees of freedom, including knee flexion/extension, internal/external rotation, adduction/abduction, anterior/posterior translation, distal/proximal translation, medial/lateral translation. The unit of angle is degree and that of translation is millimetre.
Knee flexion/extension angle at tibial vertical during gait. | 1 Day
  The gait cycle include seven key events (e.g. initial contact), and each gait has six degrees of freedom, including knee flexion/extension, internal/external rotation, adduction/abduction, anterior/posterior translation, distal/proximal translation, medial/lateral translation. The unit of angle is degree and that of translation is millimetre.
Knee adduction/abduction angle at tibial vertical during gait. | 1 Day
  The gait cycle include seven key events (e.g. initial contact), and each gait has six degrees of freedom, including knee flexion/extension, internal/external rotation, adduction/abduction, anterior/posterior translation, distal/proximal translation, medial/lateral translation. The unit of angle is degree and that of translation is millimetre.
Knee internal/external rotation angle at tibial vertical during gait. | 1 Day
  The gait cycle include seven key events (e.g. initial contact), and each gait has six degrees of freedom, including knee flexion/extension, internal/external rotation, adduction/abduction, anterior/posterior translation, distal/proximal translation, medial/lateral translation. The unit of angle is degree and that of translation is millimetre.
Knee anterior/posterior translation at tibial vertical during gait. | 1 Day
  The gait cycle include seven key events (e.g. initial contact), and each gait has six degrees of freedom, including knee flexion/extension, internal/external rotation, adduction/abduction, anterior/posterior translation, distal/proximal translation, medial/lateral translation. The unit of angle is degree and that of translation is millimetre.
Knee distal/proximal translation at tibial vertical during gait. | 1 Day
  The gait cycle include seven key events (e.g. initial contact), and each gait has six degrees of freedom, including knee flexion/extension, internal/external rotation, adduction/abduction, anterior/posterior translation, distal/proximal translation, medial/lateral translation. The unit of angle is degree and that of translation is millimetre.
Knee medial/lateral translation at tibial vertical during gait. | 1 Day
  The gait cycle include seven key events (e.g. initial contact), and each gait has six degrees of freedom, including knee flexion/extension, internal/external rotation, adduction/abduction, anterior/posterior translation, distal/proximal translation, medial/lateral translation. The unit of angle is degree and that of translation is millimetre.
Range of motion of knee flexion/extension angle | 1 Day
  The gait cycle include seven key events (e.g. initial contact), and each gait has six degrees of freedom, including knee flexion/extension, internal/external rotation, adduction/abduction, anterior/posterior translation, distal/proximal translation, medial/lateral translation. The unit of angle is degree and that of translation is millimetre.
Range of motion of knee adduction/abduction angle | 1 Day
  The gait cycle include seven key events (e.g. initial contact), and each gait has six degrees of freedom, including knee flexion/extension, internal/external rotation, adduction/abduction, anterior/posterior translation, distal/proximal translation, medial/lateral translation. The unit of angle is degree and that of translation is millimetre.
Range of motion of knee internal/external rotation angle. | 1 Day
  The gait cycle include seven key events (e.g. initial contact), and each gait has six degrees of freedom, including knee flexion/extension, internal/external rotation, adduction/abduction, anterior/posterior translation, distal/proximal translation, medial/lateral translation. The unit of angle is degree and that of translation is millimetre.
Range of motion of knee anterior/posterior translation. | 1 Day
  The gait cycle include seven key events (e.g. initial contact), and each gait has six degrees of freedom, including knee flexion/extension, internal/external rotation, adduction/abduction, anterior/posterior translation, distal/proximal translation, medial/lateral translation. The unit of angle is degree and that of translation is millimetre.
Range of motion of knee distal/proximal translation. | 1 Day
  The gait cycle include seven key events (e.g. initial contact), and each gait has six degrees of freedom, including knee flexion/extension, internal/external rotation, adduction/abduction, anterior/posterior translation, distal/proximal translation, medial/lateral translation. The unit of angle is degree and that of translation is millimetre.
Range of motion of knee medial/lateral translation. | 1 Day
  The gait cycle include seven key events (e.g. initial contact), and each gait has six degrees of freedom, including knee flexion/extension, internal/external rotation, adduction/abduction, anterior/posterior translation, distal/proximal translation, medial/lateral translation. The unit of angle is degree and that of translation is millimetre.
walking speed on the treadmill. | 1 Day

CONTACTS AND LOCATIONS:
Overall Officials: Yu Zhang, PhD, Principal Investigator — Hospital of Orthopedics, Guangzhou General Hospital of Guangzhou Military Command, 111 Liuhua Road, Guangzhou 510010, China

IPD SHARING:
Plan to Share IPD: No